CLINICAL TRIAL: NCT01541371
Title: An Open-label Prospective Trial to Explore the Tolerability, Safety and Efficacy of Flexibly Dosed Paliperidone ER in Non Acute Episode Subjects With Schizophrenia
Brief Title: A Study of Flexibly Dosed Paliperidone Extended Release Tablets in Participants With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016165; R076477-SCH-3035
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Results first posted 2013-08-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone extended-release tablets
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone ER (Experimental)
  Interventions: Drug: Paliperidone ER

INTERVENTIONS:
Drug: Paliperidone ER — Paliperidone Extended Release (ER) 3 milligram (mg) or 6 mg or 9 mg or 12 mg oral (by mouth) tablets depending on Investigator's discretion once daily for 12 weeks.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of paliperidone extended-release (ER; designed to slowly release a drug in the body over an extended period of time) tablets in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions [a false belief held in the face of strong differing evidence, especially as a symptom of psychiatric disorder] and hallucinations [imagining things], and withdrawal into the self) who were not satisfied with other prior antipsychotics (agents that control agitated psychotic behavior, alleviate acute psychotic states, reduce psychotic symptoms, and exert a quieting effect; olanzapine, quetiapine and risperidone) they had been taking. The safety and tolerability of paliperidone ER tablets will also be assessed.

DETAILED DESCRIPTION:
This is an open label (all people know the identity of the intervention), prospective (study following participants forward in time), non-randomized (the study drug is not assigned by chance, participants may choose which group they want to be in, or they may be assigned to the groups by the researchers), single-arm (getting one dose of medicine) and multi-center (when more than one hospital or medical school team work on a medical research study) study designed to determine the efficacy, tolerability and safety of flexible dosage of paliperidone ER tablets in treatment of participants with schizophrenia not satisfied with other prior antipsychotics. The duration of the study will be 12 weeks. All participants will be given paliperidone ER 3 milligram (mg) or 6 mg or 9 mg or 12 mg oral (by mouth) tablets depending on Investigator's discretion once daily for 12 weeks; initial dose for paliperidone ER will be 6 mg/day. The primary objective will be to evaluate the efficacy of treatment with paliperidone ER using Positive and Negative Symptom Scale (PANSS) total scores. Participants safety and tolerability will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants meeting Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) diagnosis criteria of schizophrenia
* Participant receiving full course of treatment (6-8 weeks) at correct dose (dose range recommended by the instruction) of Risperdal, Zyprexa or Seroquel before enrollment, was poorly controlled and had to change medication because of unsatisfying efficacy, tolerability or safety issues, or other reason
* Participant in the non-acute phase during screening received treatment with any of above three antipsychotics within 4 weeks before enrollment and state of illness was relatively stable
* 7. Female participants must be postmenopausal for at least 1 year, surgically sterile, abstinent, or, if sexually active, agree to practice an effective method of birth control before entry and throughout the study. Effective methods of birth control include prescription hormonal contraceptives, contraceptive injections, intrauterine devices, double barrier method, contraceptive patch and male partner sterilization. Female participants must also have a negative urine pregnancy test at screening
* Participant willing to and who could complete questionnaire by himself

Exclusion Criteria:

* Participant receiving treatment with clozapine or risperidone microspheres for injection (Hengde) within 3 months before screening
* Participant having history of seizure except febrile convulsion (seizures that occur during a febrile episode [fever])
* Participant having refractory schizophrenia (previous treatment with unsatisfied efficacy of 2 or more than 2 kinds of antipsychotics with different chemical structure after adequate dose and duration)
* Participant receiving electric shock treatment within 1 month before screening
* Participant having serious, unstable physical diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2008-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Janssen Pharmaceutical Ltd., China Clinical Trial, Study Director — Xian-Janssen Pharmaceutical Ltd.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 19 study centers between 30 July 2008 and 23 September 2009.
Pre-assignment Details: 405 participants were enrolled, out of which 403 participants were recruited in Safety Analysis Set (randomized and took at least 1 dose of study drug) and 394 subjects were included in full analysis set (had at least 1 efficacy evaluation).
Groups:
- Paliperidone Extended Release (ER): Paliperidone ER 3 milligram (mg) or 6 mg or 9 mg or 12 mg oral (by mouth) tablets depending on Investigator's discretion once daily for 12 weeks.
Period: Overall Study
Arm/Group | Paliperidone Extended Release (ER)
Started | 403
Full Analysis Set | 394
Completed | 326
Not Completed | 77
Not completed — Withdrawal by Subject | 14
Not completed — Lost to Follow-up | 21
Not completed — Adverse Event | 15
Not completed — Lack of Efficacy | 12
Not completed — Protocol Violation | 6
Not completed — Study medication non-compliance | 3
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Groups:
- Paliperidone Extended Release (ER): Paliperidone ER 3 milligram (mg) or 6 mg or 9 mg or 12 mg oral tablets depending on Investigator's discretion once daily for 12 weeks.
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 394
Age Continuous [Mean (Standard Deviation); unit: Years] — Information for demographics (age) was missing for 2 participants.
  Years | 30.88 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199
  Male | 195

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 12
Description: PANSS is a medical scale that assesses various symptoms of schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions [a false belief held in the face of strong differing evidence, especially as a symptom of psychiatric disorder] and hallucinations [imagining things], and withdrawal into the self). The symptoms are rated on a 7-point scale from 1 (absent) to 7 (extreme psychopathology). The total score is the sum of all 30 PANSS items, with a range of 30 (absent) to 210 (extreme ill).
Time Frame: Baseline and Week 12
Population: Full analysis set (FAS) included all participants who received at least 1 dose of study medication and had at least 1 post baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: unit on a scale
Groups:
- Lack of Efficacy Group: Paliperidone extended release (ER) tablet in flexible dose of 3, 6, 9 or 12 milligram (mg) as per Investigator's discretion was given once daily orally for 12 weeks to participants who transitioned to paliperidone ER from other oral antipsychotics for the main reason of lack of efficacy (defined as participants with a baseline total Positive and Negative Syndrome Scale [PANSS] score more than [>] or equal to [=] 70 or >=2 items scoring >=4 in the Positive or Negative Symptom Subscale or >=3 items scoring >=4 in the General Psychopathology Subscale).
- Lack of Tolerability Group: Paliperidone ER tablet in flexible dose of 3, 6, 9 or 12 mg as per Investigator's discretion was given once daily orally for 12 weeks to participants who transitioned to paliperidone ER from other oral antipsychotics for the main reason of lack of tolerability (defined as the presence of clinically relevant side effects with the previous antipsychotic medication).
- Other Group: Paliperidone ER tablet in flexible dose of 3, 6, 9 or 12 mg as per Investigator's discretion was given once daily orally for 12 weeks to participants who transitioned to paliperidone ER from other oral antipsychotics due to other reasons.
Arm/Group | Lack of Efficacy Group | Lack of Tolerability Group | Other Group
Number analyzed (Participants) | 238 | 115 | 41
unit on a scale
  Baseline | 77.18 (17.50) | 58.46 (16.31) | 63.33 (19.08)
  Change at Week 12 | -26.29 (20.77) | -13.99 (15.74) | -20.90 (18.20)

2. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Subscale Scores at Week 12
Description: PANSS is a medical scale that assesses various symptoms of schizophrenia. The symptoms are rated on a 7-point scale from 1 (absent) to 7 (extreme psychopathology). The total score is the sum of all 30 PANSS items, with a range of 30 (absent) to 210 (extreme ill). Positive syndrome subscale ranges from 7 to 49, higher change scores indicate worsening. Negative syndrome subscale ranges from 7 to 49, higher change scores indicate worsening. General Psychopathology subscale ranges from 16 to112, higher change scores indicate worsening.
Time Frame: Baseline and Week 12
Population: FAS included all participants who received at least 1 dose of study medication and had at least 1 post baseline efficacy measurement.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 394
Units on a scale
  Positive: Baseline | 17.07 (6.53)
  Positive: Change at Week 12 | -6.59 (6.30)
  Negative: Baseline | 18.57 (6.66)
  Negative: Change at Week 12 | -6.14 (5.99)
  General psychopathology: Baseline | 34.44 (9.75)
  General psychopathology: Change at Week 12 | -10.84 (10.21)

3. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Marder Subscale Scores at Week 12
Description: The PANSS is a 30-item scale to assess the neuropsychiatric symptoms of schizophrenia. The symptoms are rated on a 7-point scale from 1 (absent) to 7 (extreme psychopathology). Positive symptoms subscale consists of 8 items with total score range of 8-56; negative symptoms subscale and disorganized thoughts subscale, each consists of 7 items with total score range of 7-49, uncontrolled hostility/excitement subscale and anxiety/depression subscale, each consists of 4 items with total score range of 4-28. Higher change score indicates greater severity.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone Extended Release (ER)
Number analyzed (Participants) | 394
Units on a scale
  Positive symptoms: Baseline | 21.61 (7.15)
  Positive symptoms: Change at Week 12 | -8.16 (7.18)
  Negative symptoms: Baseline | 19.15 (7.10)
  Negative symptoms: Change at Week 12 | -6.53 (6.60)
  Disorganized thoughts: Baseline | 14.13 (4.65)
  Disorganized thoughts: Change at Week 12 | -4.13 (4.28)
  Uncontrolled hostility/excitement: Baseline | 7.73 (3.83)
  Uncontrolled hostility/excitement:Change at Week12 | -2.74 (3.63)
  Anxiety/depression: Baseline | 7.45 (2.76)
  Anxiety/depression: Change at Week 12 | -2.00 (2.67)

4. Secondary Outcome: Percentage of Participants With Response to Positive and Negative Syndrome Scale (PANSS) Total Score
Description: PANSS is a medical scale that assesses various symptoms of schizophrenia. The symptoms are rated on a 7-point scale from 1 (absent) to 7 (extreme psychopathology). The total score is the sum of all 30 PANSS items, with a range of 30 (absent) to 210 (extreme ill). Percentage of participants with at least 20 percent improvement of PANSS total score was measured.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Lack of Efficacy Group: Paliperidone ER tablet in flexible dose of 3, 6, 9 or 12 milligram (mg) as per Investigator's discretion was given once daily orally for 12 weeks to participants who transitioned to paliperidone ER from other oral antipsychotics for the main reason of lack of efficacy (defined as participants with a baseline total Positive and Negative Syndrome Scale [PANSS] score more than [>] or equal to [=] 70 or >=2 items scoring >=4 in the Positive or Negative Symptom Subscale or >=3 items scoring >=4 in the General Psychopathology Subscale).
Arm/Group | Lack of Efficacy Group | Lack of Tolerability Group | Other Group
Number analyzed (Participants) | 238 | 115 | 41
Percentage of participants | 65.97 [59.95 to 71.99] | 51.72 [42.63 to 60.82] | 61.90 [47.22 to 76.59]

5. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score at Week 12
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "normal, not at all ill" and a rating of 7 is equivalent to "among the most extremely ill participants". Higher change scores indicate worsening.
Time Frame: Baseline and Week 12
Population: FAS included all participants who received at least 1 dose of study medication and had at least 1 post baseline efficacy measurement. Here "N" (Number of Participants Analyzed): number of participants who were evaluable for this measure. 'n': number of participants who were evaluable at given time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lack of Efficacy Group | Lack of Tolerability Group | Other Group
Number analyzed (Participants) | 237 | 115 | 41
units on a scale
  Baseline (n=237,115,41) | 4.54 (0.91) | 3.20 (1.11) | 3.86 (1.09)
  Change at Week 12 (n=208,103,40) | -1.77 (0.09) | -1.01 (0.14) | -1.66 (0.23)

6. Secondary Outcome: Change From Baseline in Total Personal and Social Performance (PSP) Score at Week 12
Description: PSP assesses the degree of a participant's dysfunction within 4 domains of behavior: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior. The score ranges from 1 to 100, divided into 10 equal intervals to rate the degree of difficulty (1, absent to 6, very severe) in each of the 4 domains. Based on the four domains there will be one total score. Participants with a score of 71 to 100 have a mild degree of difficulty; from 31 to 70, varying degrees of disability; =<30, functioning so poorly as to require intensive supervision.
Time Frame: Baseline and Week 12
Population: FAS included all participants who received at least 1 dose of study medication and had at least 1 post baseline efficacy measurement. Here 'n': number of participants who were evaluable at given time point for each arm group, respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lack of Efficacy Group | Lack of Tolerability Group | Other Group
Number analyzed (Participants) | 238 | 115 | 41
Units on a scale
  Baseline (n=238,115,41) | 53.16 (13.79) | 66.95 (12.89) | 66.00 (11.21)
  Change at Week 12 (n=205,106,40) | 18.57 (16.87) | 10.09 (13.75) | 12.40 (13.33)

7. Secondary Outcome: Number of Participants With Satisfaction With the Study Treatment
Description: Participants assessed their satisfaction with paliperidone ER on a 5-point scale: 1 (very good), 2 (good), 3 (moderate), 4 (poor) and 5 (very poor).
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Lack of Efficacy Group | Lack of Tolerability Group | Other Group
Number analyzed (Participants) | 230 | 113 | 41
Participants
  Baseline, Very satisfied (n=230,113,41) | 1 | 3 | 0
  Baseline, Satisfied (n=230,113,41) | 15 | 30 | 15
  Baseline, Generally satisfied (n=230,113,41) | 84 | 58 | 25
  Baseline, Dissatisfied (n=230,113,41) | 124 | 21 | 1
  Baseline, Very dissatisfied (n=230,113,41) | 6 | 1 | 0
  Week 12, Very satisfied (n=208,105,40) | 30 | 23 | 10
  Week 12, Satisfied (n=208,105,40) | 93 | 51 | 18
  Week 12, Generally satisfied (n=208,105,40) | 62 | 24 | 10
  Week 12, Dissatisfied (n=208,105,40) | 23 | 6 | 2
  Week 12, Very dissatisfied (n=208,105,40) | 0 | 1 | 0

8. Secondary Outcome: Change From Baseline in Sleep and Daytime Drowsiness Evaluation Score at Week 12
Description: The self-administered sleep VAS scale (0-100 milimeter [mm]) rates quality of sleep (QoS) and daytime drowsiness (DD). Participants indicate mark on the scale to represent how well they have slept in the previous 7 days, score ranges from 0 mm (very badly) to 100 mm (very well); and how often they have felt drowsy within the previous 7 days, from 0 mm (not at all) to 100 mm (all the time).
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Lack of Efficacy Group | Lack of Tolerability Group | Other Group
Number analyzed (Participants) | 233 | 115 | 41
mm
  Quality of sleep score: Baseline (n=233,115,41) | 60.76 (26.70) | 75.89 (20.24) | 70.31 (22.40)
  Quality of sleep: Change at Week 12 (n=202,106,40) | 15.76 (29.46) | 2.90 (27.41) | 13.60 (26.94)
  Daytime drowsiness score: Baseline (n=233,115,41) | 38.16 (23.70) | 44.77 (25.29) | 34.26 (23.64)
  Daytime drowsiness:Change at Week 12(n=202,106,40) | -15.76 (27.52) | -21.66 (27.88) | -18.10 (26.87)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 12
Description: An undesirable or unwanted consequence that occurs during the course of the clinical trial, but not necessarily because of study drug.
Arm/Group | Paliperidone Extended Release (ER)
Serious Adverse Events (participants affected / at risk) | 1/403
Other Adverse Events (participants affected / at risk) | 227/403
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Extended Release (ER) (N=403)
Depression (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paliperidone Extended Release (ER) (N=403)
Nausea (Gastrointestinal disorders) | 15 (15)
Vomiting (Gastrointestinal disorders) | 8 (8)
Salivary hypersecretion (Gastrointestinal disorders) | 7 (8)
Constipation (Gastrointestinal disorders) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 6 (6)
Fatigue (General disorders) | 11 (14)
Hepatic function abnormal (Hepatobiliary disorders) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 15 (16)
Weight increased (Investigations) | 17 (18)
Transaminases increased (Investigations) | 9 (10)
Blood prolactin increased (Investigations) | 6 (7)
Obesity (Metabolism and nutrition disorders) | 8 (8)
Increased appetite (Metabolism and nutrition disorders) | 6 (6)
Tremor (Nervous system disorders) | 52 (56)
Dystonia (Nervous system disorders) | 35 (40)
Extrapyramidal disorder (Nervous system disorders) | 24 (28)
Dizziness (Nervous system disorders) | 17 (20)
Headache (Nervous system disorders) | 7 (9)
Akathisia (Psychiatric disorders) | 74 (76)
Somnolence (Psychiatric disorders) | 32 (33)
Insomnia (Psychiatric disorders) | 26 (28)
Sleep disorder (Psychiatric disorders) | 9 (9)
Menstrual disorders (Reproductive system and breast disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other